CLINICAL TRIAL: NCT04289597
Title: Evaluation of Difficult Airway in Obese Patients With Ultrasonography
Brief Title: Evaluation of Difficult Airway With Ultrasonography
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, Specialist Doctor-Anesthesiologist, Eskisehir Osmangazi University
Other Study IDs: ESOGU
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Difficult Intubation; Obesity
Keywords: Difficult mask; Difficult laryngoscopy; Difficult intubation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese patients: Obese patients with BMI>30
  Interventions: Diagnostic Test: Distance between hyoid bone-skin (DSHB); Diagnostic Test: Vocal cord anterior commissura-skin distance (DSAC); Diagnostic Test: minimum distance of the trachea to the skin at the level of suprasternal notch; Diagnostic Test: Thyroid isthmus-skin distance (DSI); Diagnostic Test: Skin-epiglottic distance (DSE)

INTERVENTIONS:
Diagnostic Test: Distance between hyoid bone-skin (DSHB) — Distance between hyoid bone-skin
  Other Names: DSHB
Diagnostic Test: Vocal cord anterior commissura-skin distance (DSAC) — Vocal cord anterior commissura-skin distance
  Other Names: DSAC
Diagnostic Test: minimum distance of the trachea to the skin at the level of suprasternal notch — Distance of the trachea to the skin at the level of suprasternal notch
  Other Names: DST
Diagnostic Test: Thyroid isthmus-skin distance (DSI) — Thyroid isthmus-skin distance
  Other Names: DSI
Diagnostic Test: Skin-epiglottic distance (DSE) — Skin-epiglottic distance
  Other Names: DSE

SUMMARY:
As a result of anatomical and physiological changes in obese patients, airway management can be challenging. Ultrasound measurement of neck anterior soft tissues combined with recommended predictive tests may increase the ability to predict the difficult airway. In this study we planned to evaluate the measurement of neck anterior soft tissues by ultrasound in obese patients before anesthesia induction to anticipate difficult mask ventilation, difficult laryngoscopy, and intubation.

DETAILED DESCRIPTION:
Patients with BMI> 30, schedule elective surgery under general anesthesia, and give consent will be included in the study. In the preoperative evaluation, demographic data of the patients, airway physical examination results (mouth opening, Mallampati score, thyromental distance, neck circumference (from thyroid cartilage level), abnormal upper tooth presence, neck movement restriction], presence of sleep apnea and STOP-BANG score will be recorded. In the patients taken on the operation table with supine position, ultrasound-guided soft tissue distances will be measured using ultrasound 6-13 Hz linear probe. The distance between the hyoid bone-skin (DSHB), the vocal cord anterior commissura-skin distance (DSAC), the minimum distance of the trachea to the skin at the level of the suprasternal notch (DST), the distance between the thyroid isthmus and the skin (DSI), and the distance between the epiglottis and the skin (DSE) will be measured and recorded. After standard monitoring and anesthesia induction, difficult mask ventilation will be evaluated with Han Scale [(1) can be ventilated with a mask; 2) can be ventilated with the airway (with or without muscle relaxation); 3) difficult mask ventilation (insufficient, unstable, two practitioners are needed); 4) cannot be ventilated by mask] and grade 3-4 will be recorded as difficult mask ventilation. Difficult laryngoscopy will be evaluated with Cormack Lehane Scale [grade 1: vocal cords appear; grade-2: posterior commissura and epiglottis visible; grade-3: only epiglottis are seen; grade-4: glottic structures are not visible] and grade 3-4 will be recorded as difficult laryngoscopy. Difficult intubation will also be evaluated with the number and duration of intubation attempts with the Macintosh blade. Tracheal intubation will be performed by an anesthesiologist who has at least two years of experience and unaware of ultrasound measurements. The duration of intubation (the time from the first handling of the laryngoscope until the capnography trace appeared) and the number of trials will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo general anesthesia for elective surgery
* American Anesthesiology Association physical classification (ASA) status I-III
* Body mass index (BMI) above 30

Exclusion Criteria:

* Patients with neck mass
* History of previous neck and thyroid surgery, trauma, arthritis, loss of teeth
* History of difficult intubation
* Bearded patients
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A hundred twenty-eight patients, aged 18-65 years-old, with an American Anesthesiology Association physical classification (ASA) I-III and body mass index (BMI) above 30 and planned to undergo general anesthesia for elective surgery, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Difficult Mask Ventilation | ''1 minute'' (During anesthesia induction)
  Difficult mask ventilation will be evaluated with Han scale [(1) can be ventilated with a mask; 2) can be ventilated with the airway (with or without muscle relaxation); 3) difficult mask ventilation (insufficient, unstable, two practitioners are needed); 4) cannot be ventilated by mask] and grade 3-4 will be recorded as difficult mask ventilation.

SECONDARY OUTCOMES:
Difficult laryngoscopy | ''1 minute''
  Difficult laryngoscopy will be evaluated Cormack Lehane Scale [grade 1: vocal cords appear; grade-2: posterior commissura and epiglottis visible; grade-3: only epiglottis are seen; grade-4: glottic structures are not visible] and grade 3-4 will be recorded as difficult laryngoscopy.
Difficult intubation | ''1 minute''
  Total number of intubation attempts
The duration of endotracheal intubation time | 1 minute
  The time from the first handling of the laryngoscope until the capnography trace appeared

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, MD, Principal Investigator — Teaching Assistant
Locations (1):
- Eskisehir Osmangazi Univercty, Odunpazari, Eskişehir, Turkey (Türkiye)

REFERENCES:
- [Background] Wu J, Dong J, Ding Y, Zheng J. Role of anterior neck soft tissue quantifications by ultrasound in predicting difficult laryngoscopy. Med Sci Monit. 2014 Nov 18;20:2343-50. doi: 10.12659/MSM.891037. PMID 25403231
- [Background] Ezri T, Gewurtz G, Sessler DI, Medalion B, Szmuk P, Hagberg C, Susmallian S. Prediction of difficult laryngoscopy in obese patients by ultrasound quantification of anterior neck soft tissue. Anaesthesia. 2003 Nov;58(11):1111-4. doi: 10.1046/j.1365-2044.2003.03412.x. PMID 14616599
- [Background] Liang H, Hou Y, Wei H, Feng Y. Supraglottic jet oxygenation and ventilation assisted fiberoptic intubation in a paralyzed patient with morbid obesity and obstructive sleep apnea: a case report. BMC Anesthesiol. 2019 Mar 20;19(1):40. doi: 10.1186/s12871-019-0709-7. PMID 30894124
- [Background] Murphy C, Wong DT. Airway management and oxygenation in obese patients. Can J Anaesth. 2013 Sep;60(9):929-45. doi: 10.1007/s12630-013-9991-x. Epub 2013 Jul 9. PMID 23836064
- [Background] Lundstrom LH, Moller AM, Rosenstock C, Astrup G, Wetterslev J. High body mass index is a weak predictor for difficult and failed tracheal intubation: a cohort study of 91,332 consecutive patients scheduled for direct laryngoscopy registered in the Danish Anesthesia Database. Anesthesiology. 2009 Feb;110(2):266-74. doi: 10.1097/ALN.0b013e318194cac8. PMID 19194154
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Background] Alessandri F, Antenucci G, Piervincenzi E, Buonopane C, Bellucci R, Andreoli C, Alunni Fegatelli D, Ranieri MV, Bilotta F. Ultrasound as a new tool in the assessment of airway difficulties: An observational study. Eur J Anaesthesiol. 2019 Jul;36(7):509-515. doi: 10.1097/EJA.0000000000000989. PMID 31742568